CLINICAL TRIAL: NCT06466291
Title: Registro de Enfermedad de Wilson en España
Brief Title: Spanish Wilson Disease Registry
Status: Recruiting | Type: Observational
Sponsor: Asociación Española para el Estudio del Hígado (Other)
Responsible Party: Sponsor
Other Study IDs: HCB/2021/1099
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Wilson Disease
Keywords: Genetic disease; Registry; Copper; Wilson Disease
MeSH Terms: conditions — Hepatolenticular Degeneration; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective and purpose of the Registry is to know the current status of Wilson Disease in Spain.

As secondary objectives, the prevalence and incidence of the disease will be analysed.

Likewise, the analysis aims to define future areas of interest in its pathogenesis, diagnosis, natural history, follow-up, prognosis and treatment.

Improving knowledge at a national level can help to design screening strategies and improve diagnostic circuits.

DETAILED DESCRIPTION:
Retrospective and prospective study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed Wilson Disease diagnosis

Exclusion Criteria:

* Refusal to sign the informed consent for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Wilson Disease patients under follow-up in participating centres in Spain who agree to participate in the registry by signing the informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-12-02 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
To know the current status of Wilson Disease in Spain | 2025

SECONDARY OUTCOMES:
To analyse the prevalence of Wilson Disease in Spain | 2025
To analyse the incidence of Wilson Disease in Spain | 2025

OTHER OUTCOMES:
To define future areas of interest in Wilson Disease | 2025
  To define future areas of interest in the disease pathogenesis, diagnosis, natural history, follow-up, prognosis and treatment

CONTACTS AND LOCATIONS:
Overall Officials: Zoe Mariño, Study Director — Asociación Española para el Estudio del Hígado
Locations (1):
- Hospital Clinic, Barcelona, Spain